CLINICAL TRIAL: NCT02914301
Title: Effectiveness of a Mobile App for Prenatal Care to Safely Reduce In-Person Visits and Improve Patient Satisfaction: Study Protocol for a Multicenter Prospective Quasi-Randomized Trial
Brief Title: Mobile App for Prenatal Care to Reduce Visits and Improve Satisfaction Study
Acronym: SPROUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew Meltzer (Other)
Collaborators: 1EQ, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Andrew Meltzer, Principal Investigator, George Washington University
Organization: George Washington University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BABYSCRIPTS 1B
Record Dates: First submitted 2016-09-08; First posted 2016-09-26 (Estimated); Results first posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-11

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Babyscripts Prenatal App (Active Comparator): For patients allocated to the experimental group, they will be assisted in downloading the BRx app to their smartphone and set up the connected weight scale and blood pressure cuff. At time of enrollment, research assistant will also collect baseline demographic and clinical data. For patients allocated to this study arm, the clinician will be informed and therefore, will be receiving regular app-based education while the clinician will be receiving regular blood pressure and weight measurements. Following that communication, it will be the physicians' judgement to reduce in-person visits from usual care.
  Interventions: Device: Babyscripts Prenatal App
- Placebo (Placebo Comparator): For patients cared for by clinicians allocated to the control (usual care) arm, the clinician will discuss the management options and scheduling procedures with the patient in that clinician's usual fashion. The patient will not be given access to the BRx app but will consent to the study data collection and survey administration. All potential study subjects will receive standard medical care per DoD/VA Clinical Practice Guidelines for Management of the uncomplicated pregnancy (REF) and local preference by board-certified OB/GYN physicians.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Babyscripts Prenatal App — The use of a mobile digital app to facilitate certain aspects of standard prenatal care.
  Arms: Babyscripts Prenatal App
Device: Placebo — No Mobile App, Usual care
  Arms: Placebo

SUMMARY:
Prenatal care is defined as preventive healthcare characterized by regular check-ups by doctors or midwives to treat and prevent potential health problems throughout the course of the pregnancy. The investigators propose that a mobile app for prenatal care has the potential to provide patient-tailored, risk-appropriate prenatal educational content and may facilitate vital sign and weight checks between visits. The investigators describe the methods used to develop and test the effectiveness of a mobile app for prenatal care to safely reduce the number of in-person visits to the obstetrician (OB) compared to standard of care.

DETAILED DESCRIPTION:
This is a protocol for a multi-center quasi-randomized controlled trial to compare an intervention group receiving a prenatal care app, to a control group receiving usual care. The trial is being conducted at two diverse outpatient obstetric practices that are part of a single academic department of obstetrics in Washington, DC. Women who are between 18 and 40, who are visiting their OB for a first trimester routine visit, who have a confirmed desired pregnancy, who are not considered "high-risk," and who have an IOS, Android or Windows-based smart phone that they use regularly will be eligible for enrollment. The Investigators will measure the effect of a mobile app for prenatal care on:

1. the number of in-person OB visits during pregnancy;
2. patient satisfaction with prenatal care;
3. gestational weight gain;
4. maternal and fetal outcomes; and
5. clinician satisfaction.

To capture these outcomes, the investigators will administer patient surveys via telephone every 4 weeks during gestation and the immediate post-partum period, review the electronic medical record, and conduct in-depth interviews with a representative subset of patients after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be women who are between 18 than 40-years-old, who are visiting the OB for a first-trimester verification of pregnancy visit, new OB visit or follow-up OB visit, who are low-risk per treating OB, who regularly use a smart-phone, who can understand and consent to English-written consent form.
* Eligible clinicians will be attending obstetric physicians who refer the patient to the research assistant for informed consent and full eligibility assessment.

Exclusion Criteria:

* High-risk obstetrical condition*
* Intends midwifery care
* Intends to terminate
* Not Local resident
* Non--English speaker

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew C Meltzer, MD, MS, Principal Investigator — The George Washington University
Locations (1):
- George Washington University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marko KI, Ganju N, Krapf JM, Gaba ND, Brown JA, Benham JJ, Oh J, Richards LM, Meltzer AC. A Mobile Prenatal Care App to Reduce In-Person Visits: Prospective Controlled Trial. JMIR Mhealth Uhealth. 2019 May 1;7(5):e10520. doi: 10.2196/10520. PMID 31042154
- See also: site for mobile app — https://getbabyscripts.com/
- Available data/document: Informed Consent Form: FWA00005945 — https://files.acrobat.com/a/preview/c262292c-6de1-4f73-bae3-689555b8c77f
- Available data/document: Individual Participant Data Set: Post-Partum Survey — https://files.acrobat.com/a/preview/5ec925dd-52ad-4b07-b6fc-2084d2f751d5
- Available data/document: Individual Participant Data Set: Prenatal Participant Data -22 — https://files.acrobat.com/a/preview/984213bb-ccef-419b-8f56-87336004ec5a

RESULTS

PARTICIPANT FLOW:
Groups:
- Babyscripts Prenatal App: For patients allocated to the study group, they will be assisted in downloading the BRx app to their smartphone and set up the connected weight scale and blood pressure cuff. At time of enrollment, research assistant will also collect baseline demographic and clinical data. For patients who were allocated to the intervention arm, the clinician will told that they are in intervention group and therefore will be receiving regular app-based education and clinician will be receiving regular blood pressure and weight measurements. Following that communication, it will be the physicians' judgement to reduce in-person visits from usual care.
  Babyscripts Prenatal App: The use of a mobile digital app to facilitate certain aspects of standard prenatal care.
- Placebo: For patients cared for by clinicians allocated to the usual care arm, the clinician will discuss the management options and scheduling procedures with the parent in that clinician's usual fashion. The patient will not be given access to the BRx app but will consent to the study data collection and survey administration. All potential study subjects will receive standard medical care per DoD/VA Clinical Practice Guidelines for Management of the uncomplicated pregnancy (REF) and local preference by board-certified OB/GYN physicians.
  Placebo: No Mobile App, Usual care
Period: Overall Study
Arm/Group | Babyscripts Prenatal App | Placebo
Started | 60 | 58
Completed | 47 | 41
Not Completed | 13 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Babyscripts Prenatal App | Placebo | Total
Number analyzed (Participants) | 47 | 41 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.0 (3.3) | 32.2 (3.2) | 32.6 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 41 | 88
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American | 14 | 13 | 27
  Other | 33 | 28 | 61
Region of Enrollment [Number; unit: participants]
  United States | 47 | 41 | 88
College Graduate [Count of Participants; unit: Participants] | 45 | 36 | 81
Gravidity Per Patient [Count of Participants; unit: Participants]
  One | 25 | 22 | 47
  Greater than One | 22 | 19 | 41
Parity Per Patient [Count of Participants; unit: Participants]
  Zero | 30 | 25 | 55
  Greater than One | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Total Visit Number
Description: In discussions with OBs, it became clear that, patient safety notwithstanding, the advantages and disadvantages of a reduced visit schedule versus usual care were of greatest importance and so total visit number was selected as the primary outcome. We will measure total visit number by reviewing the EHR. All other outcomes will be secondary outcomes.
Time Frame: From first trimester up to postpartum, between 6 and 9 months
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Babyscripts Prenatal App | Placebo
Number analyzed (Participants) | 45 | 51
visits | 7.9 (1.8) | 10.2 (1.8)
Statistical Analysis 1: Comparison: Babyscripts Prenatal App vs Placebo; Test type: Other — We compared outcomes between study arms using t-tests for continuous outcomes; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Gestational Weight Gain
Description: We will assess gestational weight gain following enrollment until delivery. These measures will be obtained by health record review and review of data collected in the app. Data collection will be performed with a standardized data collection sheet and a 10% check for interrater reliability.
Time Frame: From first trimester up to postpartum, between 6 and 9 months
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Babyscripts Prenatal App | Placebo
Number analyzed (Participants) | 45 | 51
pounds
  Underweight (BMI< 18.5) | 22.9 (13.4) | 20.9 (4.8)
  Normal (18.5<BMI<25) | 34.0 (8.4) | 30.5 (7.7)
  Overweight (25<BMI<30) | 35.0 (10.8) | 24.2 (11.2)
  Obese (BMI>30) | 13.0 (0) | 9.4 (9.6)

ADVERSE EVENTS:
Arm/Group | Babyscripts Prenatal App | Placebo
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/51
Other Adverse Events (participants affected / at risk) | 0/45 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No